CLINICAL TRIAL: NCT03545581
Title: Metabolic Effects of Short-term Dietary Supplementation With Fructose in Carriers for Hereditary Fructose Intolerance
Brief Title: Fructose Supplementation in Carriers for Hereditary Fructose Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: University of Liege (Other)
Responsible Party: Principal Investigator, Christel Tran, Principal Investigator, University of Lausanne
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2016-00289
Record Dates: First submitted 2018-05-07; First posted 2018-06-04 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Hereditary Fructose Intolerance
Keywords: Fructose; Uric acid; Glucose homeostasis
MeSH Terms: conditions — Fructose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental diet Fru rich diet (Other): Enriched fructose diet from day 1 to day 7.
  Interventions: Other: Experimental diet Fru rich diet
- Experimental low Fru diet (Other): Low fructose diet from day 1 to day 7.
  Interventions: Other: Experimental low Fru diet

INTERVENTIONS:
Other: Experimental diet Fru rich diet — 7 days (day 1 to day 7) with fructose enriched drinks 3x/d. Test meal at day 7 with fructose (0.7 g/body weight) and glucose (0.7 g/body weight)
  Arms: Experimental diet Fru rich diet
Other: Experimental low Fru diet — 7 days (day 1 to day 7) with low-fructose diet (<10g/d). Test meal at day 7 with fructose (0.7 g/body weight) and glucose (0.7 g/body weight)
  Arms: Experimental low Fru diet

SUMMARY:
This study aimed to examine metabolic response to a short-term fructose enriched diet in carriers for hereditary fructose intolerance compared to controls. Effects of fructose coffees will be assessed in 7 healthy volunteers and 7 subjects with heterozygous mutation for ALDOB gene in a randomized, controlled, crossover trial.

DETAILED DESCRIPTION:
A high fructose intake also increases blood lactate and uric acid concentrations. It has been proposed that uric acid may contribute to insulin resistance by impairing endothelium-dependent vasodilation, promoting pro-inflammatory effects and dyslipidemia by activating de novo lipogenesis.

These consequences of fructose overconsumption may be even more marked in individuals with hereditary alterations in fructose metabolism. Indeed, individuals with hereditary fructose intolerance (HFI), due to biallelic mutations in the gene coding for aldolase B (ALDOB), may develop acute, life-threatening manifestations when exposed to fructose. Heterozygous carriers of ALDOB mutation are quite common in the general population, with a predicted frequency ranging between 1:55 and 1:120. Few studies have examined the effect of fructose ingestion in heterozygotes subject for HFI. Heterozygous carriers are generally considered to have normal fructose metabolism since a ~ 50% level of aldolase B activity is presumed to be sufficient for adequate function. However, heterozygous carriers were reported to have enhanced uric acid responses to large intravenous and/or oral fructose loads.

Investigators hypothesized that heterozygous carriers may also have mild defects of fructose metabolism and/or a larger increase in cardiometabolic risk factors than the normal population after ingestion of moderate amounts of fructose.

ELIGIBILITY:
Inclusion Criteria:

* Case subjects: Heterozygous carriers for ALDOB mutation confirmed by molecular analysis
* Control subjects: healthy individuals matched for weight and age to subjects

Exclusion Criteria:

* Fasting glucose > 7.0 mmol/L
* Fasting triglycerides > 4.0 mmol/L
* Chronic renal insufficiency (eGFR < 50 ml/min)
* Drugs
* Women who are pregnant or breast feeding
* For women: lack of safe contraception
* Alcool consumption > 30g/d
* Inability to discern

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Metabolite concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  The primary endpoint is the change of metabolite concentration after ingestion of a test meal (oral glucose and fructose load) under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design

SECONDARY OUTCOMES:
Plasma glucose concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in glucose concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma insulin concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in insulin concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma fructose concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in fructose concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma uric acid concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in uric acid concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma lactate concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in lactate concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma urea concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in urea concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma creatinine concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in creatinine concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma phosphate concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in phosphate concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma triglycerides concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in triglycerides concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma metabolome concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in metabolome concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma ammonia concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in ammonia concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma amino acid concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in amino acid concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma alanine transaminase (ALAT) concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in alanine transminase (ALAT) concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Plasma aspartate transaminase (ASAT) concentration | Time Frame: -30 min before ingestion of a test meal to 120 min after ingestion of a test meal
  Change in aspartate transaminase (ASAT) concentration after ingestion of a test meal under 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
Urine metabolome concentration | Time Frame: 24 hour urine collection before ingestion of a test meal and after 7 days of 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
  Change in urine metabolome profile after low fructose diet and an enriched fructose diet according to a crossover design
Urine creatinine concentration | Time Frame: 24 hour urine collection before ingestion of a test meal and after 7 days of 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
  Change in urine creatinine profile after low fructose diet and an enriched fructose diet according to a crossover design
Urine urea concentration | Time Frame: 24 hour urine collection before ingestion of a test meal and after 7 days of 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
  Change in urine urea profile after low fructose diet and an enriched fructose diet according to a crossover design
Urine uric acid concentration | Time Frame: 24 hour urine collection before ingestion of a test meal and after 7 days of 2 conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
  Change in urine uric acid profile after low fructose diet and an enriched fructose diet according to a crossover design
Body weight | Time Frame: at baseline before study intervention and at the end of each conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
  Change of body weight after low fructose diet and an enriched fructose diet according to a crossover design
Blood pressure | Time Frame: at baseline before study intervention and at the end of each conditions (enriched fructose diet vs poor fructose diet) according to a crossover design
  Change of systolic and diastolic pressure after low fructose diet and an enriched fructose diet according to a crossover design

CONTACTS AND LOCATIONS:
Locations (1):
- Guillaume Debray, Liège, Belgium

REFERENCES:
- [Derived] Debray FG, Seyssel K, Fadeur M, Tappy L, Paquot N, Tran C. Effect of a high fructose diet on metabolic parameters in carriers for hereditary fructose intolerance. Clin Nutr. 2021 Jun;40(6):4246-4254. doi: 10.1016/j.clnu.2021.01.026. Epub 2021 Jan 27. PMID 33551217